CLINICAL TRIAL: NCT06106360
Title: A Pilot Prospective Clinical Trial Using Remote Patient Monitoring for Cancer Patients Undergoing Outpatient Chemotherapy
Brief Title: A Pilot Prospective Clinical Trial Using Remote Monitoring for Cancer Patients Undergoing Outpatient Chemotherapy
Status: Recruiting | Type: Observational
Sponsor: Inova Health Care Services (Other)
Responsible Party: Sponsor
Other Study IDs: U23-08-5132
Record Dates: First submitted 2023-10-24; First posted 2023-10-30 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Solid Tumor; Hematological Malignancy
Keywords: Wearable Electronic Devices
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 120 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (1):
- 3 Cohorts: Cohort 1: Daily from day 2 through the end of treatment cycle (n=34) Cohort 2: Daily days 2-9 then every third day through end of cycle (n=33) Cohort 3: Daily days 2-9 for all symptoms, every third day thereafter regarding 'pain' only through end of cycle (n=33)
  Interventions: Device: Locus Health iPhone App

INTERVENTIONS:
Device: Locus Health iPhone App — In this pilot study patients are enrolled into three (3) different groups which will vary by the frequency of the queries being sent to the patients during their chemotherapy cycle. The patients will be separated into three groups of 33-34 patients each. Each group will have a different frequency of symptom questions sent to them via the Locus Health iPhone App to determine patient fatigue and the compliance impact of different query cadences. Patients will be assigned to these 3 groups sequentially since the platform could not assign patients to these three cohorts in a random manner.

SUMMARY:
A pilot study using remote monitoring technology developed by Locus Health in cancer patients undergoing chemotherapy treatment.

DETAILED DESCRIPTION:
Modern-day wearable devices, such as Apple Watches or Fitbits, are widely available, non-invasive, and can provide continuous vital sign monitoring for the early detection of potential health complications. Early detection of things such as fever or increased heart rate can alert patients to seek medical attention sooner and therefore have the potential to improve patient outcomes and decrease healthcare costs.

To further investigate the feasibility of using remote patient monitoring ( RPM)to prospectively monitor patients undergoing outpatient chemotherapy for chemotherapy related toxicities, defined as follows: (1) patients answer queries through the Locus Health iPhone app at least 70% of the time; (2) patients report that the Locus Health iPhone app and the Apple Watch were 'easy to use,' defined as an average score of 7 or higher on the first two questions of the post-intervention questionnaire, and (3) fewer than 10% of patients withdraw from the study.

ELIGIBILITY:
Inclusion Criteria:

* Planned to be treated with a new cytotoxic chemotherapy or chemoimmunotherapy regimen for a solid tumor or malignant hematology condition for at least 4 months
* ECOG performance status of 0-2
* Age of 18 or older patient with any solid tumor or hematologic malignancy
* English or Spanish speaker
* Own an Apple iPhone
* Capacity and willingness to provide informed consent

Exclusion Criteria:

* Patients undergoing concurrent radiation since they will be seen on a daily basis by clinic care teams and are not likely to benefit from active remote patient monitoring
* Patients unwilling or unable to comply with the protocol, including wearing the Apple Watch (including recharging daily) and answering queries on the Locus Health iPhone application per the protocol and study group cadence
* Any condition for which in the Investigator's opinion would limit compliance with study requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a wide range of solid tumor and malignant hematology malignancies will be enrolled
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-10-26 (Actual); Primary Completion 2025-11-01 (Actual); Study Completion 2026-06-26 (Estimated)

PRIMARY OUTCOMES:
The Use of Locus Heath iPhone App and the Apple Watch by Participants Undergoing Outpatient Chemotherapy. | 120 days or until the chemotherapy regimen has stopped, whichever is sooner
  The feasibility is determined when 80% of the patients wear the watch at least 70% of the time during waking hours.

CONTACTS AND LOCATIONS:
Overall Officials: John Deeken, MD, Principal Investigator — Inova Schar Cancer Institute
Locations (1):
- Inova Schar Cancer Institute, Fairfax, Virginia, United States

IPD SHARING:
Plan to Share IPD: Yes
* Age, gender, race/ethnicity
  * Active Problem List
  * Past Medical History
  * Past Surgical History
  * Social History
  * Vital Measurements from each clinic visit
  * Lab Results
  * Medication Orders
  If the patient is seen in the Emergency Room or hospitalized, the following data will be extracted:
  * ER/Hospital Based Problem List
  * ER/ Hospital reason for presentation/Admission
  * Hospital Admission Diagnoses
Supporting Information: CSR
Time Frame: The Apple/Locus Health RPM intervention will end and the patient will come off study when the chemotherapy regimen is stopped for any reason.
Access Criteria: All patient records and end-of study questionnaires will be de-identified using a letter and number assigned to their case at the time of enrollment on study. No record used for the data analysis will contain information which could identify the patient. Only the delegated research team will have access to the 'key' which connects patient identifiable information with this assigned number For computer records, the key will be protected by a double-password protection system. Any paper records will be contained in a locked cabinet within a locked office to ensure patients' privacy is protected.

REFERENCES:
- [Result] Heinz WJ, Buchheidt D, Christopeit M, von Lilienfeld-Toal M, Cornely OA, Einsele H, Karthaus M, Link H, Mahlberg R, Neumann S, Ostermann H, Penack O, Ruhnke M, Sandherr M, Schiel X, Vehreschild JJ, Weissinger F, Maschmeyer G. Diagnosis and empirical treatment of fever of unknown origin (FUO) in adult neutropenic patients: guidelines of the Infectious Diseases Working Party (AGIHO) of the German Society of Hematology and Medical Oncology (DGHO). Ann Hematol. 2017 Nov;96(11):1775-1792. doi: 10.1007/s00277-017-3098-3. Epub 2017 Aug 30. PMID 28856437
- [Result] Kuderer NM, Dale DC, Crawford J, Cosler LE, Lyman GH. Mortality, morbidity, and cost associated with febrile neutropenia in adult cancer patients. Cancer. 2006 May 15;106(10):2258-66. doi: 10.1002/cncr.21847. PMID 16575919
- [Result] Zimmer AJ, Freifeld AG. Optimal Management of Neutropenic Fever in Patients With Cancer. J Oncol Pract. 2019 Jan;15(1):19-24. doi: 10.1200/JOP.18.00269. PMID 30629902
- [Result] Verma N, Haji-Abolhassani I, Ganesh S, Vera-Aguilera J, Paludo J, Heitz R, Markovic SN, Kulig K, Ghoreyshi A. A Novel Wearable Device for Continuous Temperature Monitoring & Fever Detection. IEEE J Transl Eng Health Med. 2021 Jul 19;9:2700407. doi: 10.1109/JTEHM.2021.3098127. eCollection 2021. PMID 34765323